CLINICAL TRIAL: NCT01175005
Title: Procalcitonin as a Marker of Serious Infection in Patients With Fever and a Central Venous Catheter
Brief Title: Procalcitonin Levels in Patients With Fever and a Central Line
Status: Completed | Type: Observational
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Amanda Kasem, MD Principal Investigator, Phoenix Children's Hospital
Other Study IDs: PCH 10-042
Record Dates: First submitted 2010-07-28; First posted 2010-08-04 (Estimated); Results first posted 2011-04-27 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Fever
Keywords: Fever; Central venous catheter; Procalcitonin; Fever with a central venous catheter
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Fever and a central venous catheter

SUMMARY:
Procalcitonin (PCT) is one of many inflammatory markers which rises in response to infection. Many studies have shown this marker to be more indicative of a patient's clinical course in comparison to other inflammatory markers, such as Erythrocyte Sedimentation Rate (ESR) and C reactive protein (CRP), when assessing a patient's risk for serious infection. A particular population with potential for serious infection is that of the patient with fever and a central line, most often secondary to an oncologic disease. These patients are often neutropenic and unable to fight off infection, thereby rendering them extremely vulnerable to rapid declines in clinical status. By identifying a level of procalcitonin which is significant as a threshold for serious bacterial infection, the investigators can very early on identify the sickest patients and those who could potentially have a worse clinical course and/or outcome.

The primary study goal is to identify whether a level of procalcitonin exists above which rates of bacteremia or serious bacterial infections in patients with fever and a central line exist. The investigators will try to determine if levels of PCT correlate with bacterial infection in line sepsis in the specific population of patients who most often have a central line secondary to an oncologic process. The investigators proposed this theory since peak values of PCT have been shown to be elevated in acute settings making it a useful tool in this particular population.

DETAILED DESCRIPTION:
A prospective study in which patients presenting to the Emergency Department (ED) with fever and a central line will have procalcitonin levels checked, along with their CBC and blood culture. Procalcitonin levels will be recorded and blood culture results will be followed to see whether higher procalcitonin levels correlate with a greater risk of having a positive blood culture.

A prospective study will be conducted on patients with fever and a central line who present to the Emergency Department. Written informed consent will be obtained for each patient. We will include all patients 18 years of age and younger and exclude patients who had received antibiotics within the previous 24 hours of presenting to the ED as studies have shown that PCT levels dramatically decrease with the institution of antibiotic therapy. Patients will be identified on presentation to our ED with a chief complaint of "Fever and Central Venous Catheter". Diagnosis of sepsis will be made by clinical findings (fever, chills, altered mental status…) and confirmed by laboratory findings (leukocytosis or leucopenia with neutropenia, and later positive blood cultures). Management of each individual patient was determined by the pediatric emergency medicine physician in consult with a pediatric hematologist-oncologist and, in required cases, by an intensivist.

On presentation to the ED, all patients will have a CBC with differential, blood culture from the central line and procalcitonin levels drawn. All will receive empiric antibiotics initiated with either Ceftriaxone (if the patients is clinically stable and non-neutropenic defined as an Absolute Neutrophil Count (ANC)>1500 cells/microliter) or with Cefepime and Gentamicin in the neutropenic or ill appearing patient.

Electronic medical records will be reviewed for patient demographics, medical and social history and clinical presentation. Medical records during admission will be used to follow the progression and hospital stay as well as the management used. Office records will be used for post admission outcomes.

Levels of PCT will be determined using the Brahms Kryptor compact which required a minimum of 200 microliters of plasma, serum or whole blood to run a PCT level and could detect a level as low as <0.02ng/ml within 20-25 minutes. Levels reported as <0.05ng/ml are considered not indicative of sepsis while levels >2 ng/ml are indicative of high sepsis probability. Levels in between 0.05 and 2 suggest a repeat level be drawn after 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and younger
* Fever and a central venous catheter
* Presentation to an Emergency Department
* Central line secondary to Hematologic/Oncologic, Renal or Gastrointestinal disease

Exclusion Criteria:

* Intravenous antibiotics in the 24 hours prior to presentation
* PICC line
* Parental refusal or inability to provide consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with fever and a central venous catheter who are 18 years of age and younger will be enrolled and will have PCT levels drawn in the Emergency Department.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Kasem, MD, Principal Investigator — Phoenix Children's Hospital

REFERENCES:
- [Derived] Kasem AJ, Bulloch B, Henry M, Shah K, Dalton H. Procalcitonin as a marker of bacteremia in children with fever and a central venous catheter presenting to the emergency department. Pediatr Emerg Care. 2012 Oct;28(10):1017-21. doi: 10.1097/PEC.0b013e31826caac2. PMID 23023470

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fever and a Central Venous Catheter
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fever and a Central Venous Catheter
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 62
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 6 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 62
Neutropenic [Number; unit: participants] — Number of patients who were neutropenic defined as ANC less than 1500 cells/microliter
  participants
    neutropenic | 27
    Non neutropenic | 35
Blood culture [Number; unit: participants] — Blood culture negative vs positive
  participants
    Blood culture negative | 48
    Blood culture positive | 14

OUTCOME MEASURES:

1. Primary Outcome: Procalcitonin Level at ED Presentation
Description: Level of procalcitonin will be obtained. At the end of the study we will determine who was septic or bacteremic and compare the procalcitonin levels between those who were septic/bacteremic and those who were not.We will attempt to identify whether a level of procalcitonin exists above which rates of bacteremia or bacterial sepsis in patients with fever and a central line exist. Blood cultures will be followed for up to 5 days until reported as final.There are no further study interventions.
Time Frame: Initial blood draw in ED and if admitted a second level will be obtained at 24 hours.
Measure: Mean (95% Confidence Interval); unit: ng/dL
Groups:
- Blood Culture Positive: Procalcitonin level in patients with fever and a CVC with positive blood culture
- Blood Culture Negative: Procalcitonin level in patients with fever and a CVC with negative blood culture
Arm/Group | Blood Culture Positive | Blood Culture Negative
Number analyzed (Participants) | 14 | 48
ng/dL | 18.47 [17.42 to 19.52] | 0.65 [0.08 to 1.22]
Statistical Analysis 1: Comparison: Blood Culture Positive vs Blood Culture Negative; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Fever and a Central Venous Catheter
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes